CLINICAL TRIAL: NCT00687115
Title: Predicting Adaptive Thermogenesis
Brief Title: Predicting Weight Gain and Weight Loss Associated With Overeating or Fasting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 999908140; 08-DK-N140
Record Dates: First submitted 2008-05-29; First posted 2008-05-30 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-10-06

CONDITIONS: Obesity; Diet Therapy; Weight Loss; Weight Gain; Nutrition Therapy
Keywords: 24 Hour Energy Expenditure; Respiratory Chamber; Obesity; Weight Loss; Overfeeding
MeSH Terms: conditions — Obesity; Weight Loss; Weight Gain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Overfeeding (Other): an inpatient overfeeding arm in which obesity resistant individuals are prescribed a 150% increase in a weight maintenance calorie diet for 6 weeks which (by random assignment) is either low in protein (6%) content. Overfeeding or Overfeeding Low Pro or with normal (20%) protein content
  Interventions: Behavioral: Overfeeding; Behavioral: Overfeeding Low Pro
- Weight Loss (Other): a weight loss arm in which obese individuals are placed on a 50% decrease from a weight maintenance calorie diet for 6 weeks which (by random assignment) is either a standard 50% decrease in energy intake with all macronutrients held at the same percentage (20% protein, 50% carbohydrate, 30% fat) or a 50% decrease in energy intake with the same absolute protein content (in grams) as the weight maintaining diet while on our clinical research unit then followed as outpatients monthly for 10 months
  Interventions: Behavioral: Weight Loss

INTERVENTIONS:
Behavioral: Weight Loss — liquid diet at 50% of weight maintaining intake
  Arms: Weight Loss
Behavioral: Overfeeding — Overfeeding at 150% of weight maintaining intake
  Arms: Overfeeding
Behavioral: Overfeeding Low Pro — Overfeeding 150% of normal intake at <5% protein
  Arms: Overfeeding

SUMMARY:
This study will investigate how to better predict why some individuals gain or lose weight more easily than others. It will examine whether the increase in the amount of energy a body burns in 24 hours with overeating or the decrease over 24 hours with fasting can help determine how easily someone gains or loses weight.

Healthy people between 18 and 60 years of age who have a body mass index (BMI) between 18.5 kg/m(2) and 24 kg/m(2) (for overfeeding study) or a BMI greater than 27 kg/m(2) with a body weight less than 350 pounds (weight loss study) may be eligible for this study. The study requires a 10-week admission to the NIH Clinical Center (2-week baseline, 6-week overfeeding/weight loss, 2-week post-weight change).

Participants undergo the following tests and procedures during the hospital admission:

* Medical history, physical examination and laboratory studies
* Questionnaires to assess eating behavior, food preferences, body composition, and activity level
* Body composition assessment (height, weight, waist circumference, and fat mass and muscle content through DXA and MRI scans)
* Oral glucose tolerance test
* Meal test to measure the response of certain hormones to food
* Activity monitors to determine activity level
* Metabolic chamber study to measure calories burned over 24 hours and monitor body temperature
* Free-living energy use study to measure calories burned under normal home conditions over 7 days
* Fat and muscle biopsies
* Dietary intervention: Measurements of food intake and energy loss over a 6-week overfeeding (1.5 times the subject s normal food intake) or weight loss (one-half the subject s normal food intake) program

Followup procedures after the inpatient stay:

* Height and weight measurements at 6 months (overfeeding study participants) and monthly for the first year, at 3-month intervals for the second year, and then yearly for 3 more years (weight loss study participants)
* Yearly visits (2-night inpatient stay) for all participants for repeat meal test, DXA, oral glucose tolerance test, behavioral questionnaires and, in women who can become pregnant, pregnancy test

DETAILED DESCRIPTION:
For obese individuals, losing weight and keeping it off are extremely difficult, whereas some other individuals are thin and report trouble gaining weight. In most weight loss and overfeeding studies there is a large variation in the amount of weight lost or gained, and it is not clear whether an individual s response to an intervention can be predicted. Measurement of the amount of energy an individual uses over 24 hours (24 hour energy expenditure or 24-EE) and the response of 24-EE to overfeeding and fasting may help predict which individuals will have the greatest changes in weight with changes in energy balance. In previous work, 24-EE responses to overfeeding and fasting were related such that individuals with the greatest increase in 24-EE upon overfeeding tended to have the smallest decrease in 24-EE upon fasting ( spendthrift phenotype) and those individuals with less increase in 24-EE during overfeeding had a greater decrease in 24-EE with fasting ( thrifty phenotype). Those with the spendthrift phenotype who had a greater increase in 24-EE in response to overfeeding gained less weight over time. Furthermore, studies have shown that diets with very low protein content may magnify the variability in response to overfeeding.

The aim of this study is to determine if a phenotype defined by 24-EE responses to overfeeding and underfeeding is related to weight loss or gain in 4 different under- and overfeeding settings: an inpatient weight loss group for obese individuals who will be administered one of two diets based on a 50% reduction of their daily energy needs for six weeks (standard reduction diet or calorie reduced diet that is still high in protein; 6 week weight reduction, 10 week stay, n=20/standard reduction diet group and n=10/relative high protein diet), and two overfeeding groups for lean, weight gain resistant individuals: a low-protein overfeeding group at 150% of daily energy needs for 6 weeks overfeeding (6% protein, 64% carbohydrate, 30% fat; 10 week stay, n=10), and a normal protein overfeeding group at 150% of daily energy needs for 6 weeks overfeeding (20% protein, 50% carbohydrate, 30% fat; 10 week stay, n=10). We will also examine additional metabolic and behavioral measurements to determine how they relate to weight change and changes in 24-EE. These include sympathetic nervous system activity, behavior, adipose and muscle tissue energy content, and abdominal adipocyte size. The study will evaluate the relationship between the percent increase in 24-EE in response to overfeeding/underfeeding and the amount of weight change over time in each subject. These findings may provide important information for predicting and adapting specific individualized interventions for obesity.

ELIGIBILITY:
* INCLUSION CRITERIA:
* BMI greater than or equal to 27 kg/m(2) for the weight loss protocol but body weight less than 350 pounds to accommodate the DXA scanner.
* BMI less than or equal to 24 kg/m(2) (and BMI greater than or equal to 18.5 kg/m(2) for the overfeeding protocols. A history of low BMI and difficulty gaining weight.
* Age 18-60 years, to minimize potential co-morbid conditions which may indirectly affect EE. Minors under the age of 18 will be excluded because growth and pubertal issues are significant parameters that could affect our outcomes and also because the time requirements of the study are such that they would interfere with school schedules. Women who are post-menopausal will be excluded from the study as changes in their metabolism could affect the baseline measurements which are hypothesized to predict weight change.
* Healthy, as determined by medical history, physical examination, and laboratory tests

EXCLUSION CRITERIA:

* Current smoking
* Type 2 diabetes (according to the World Health Organization diagnostic criteria)
* Impaired glucose tolerance (according to the World Health Organization diagnostic criteria) for those participating in the overfeeding study arms only
* Endocrine disorders (Cushing s Disease, pituitary disorders, and hypo- and hyperthyroidism)
* Chronic pulmonary disorders, including chronic obstructive pulmonary disease that would limit ability to follow the protocol (investigator judgment) and obstructive sleep apnea syndrome; only subjects with mild or exercise-induced asthma on no medications or on beta-adrenergic agonists only (such as albuterol) will be allowed to enter the study (provided use of these agents is not required for one week before study entry).
* Cardiovascular diseases (coronary heart disease, heart failure, arrhythmias, and peripheral artery disease)
* Hypertension (blood pressure measurement higher than 140/90 mm Hg (overfeeding study) or 160/95 (weight loss study) on two or more occasions or use of anti-hypertensive medications)
* Diagnosed gastrointestinal diseases, including inflammatory bowel diseases (e.g., Crohn s disease and ulcerative colitis), malabsorption syndromes (e.g., celiac disease), gastric ulcer (active); only subjects with gastro-esophageal reflux will be allowed to enter the study
* Presence of a pacemaker or other implantable devices/shrapnel which may interfere with the MRI or CorTemp measurements
* Liver disease (cirrhosis, active hepatitis B or C, and AST or ALT greater than or equal to 1.5 times normal)
* Renal disease (serum creatinine concentrations greater than or equal to 1.5 mg/dl and/or overt proteinuria)
* Central nervous system disease (cerebrovascular accidents, dementia, and neurodegenerative disorders)
* Cancer requiring treatment in the past five years, except for non-melanoma skin cancers or cancers that have clearly been cured or in the opinion of the investigator carry an excellent prognosis (e.g., Stage 1 cervical cancer)
* Alcohol (more than 3 drinks per day) and/or drug abuse (such as amphetamines, cocaine, heroin, or marijuana)
* Current or past history of: bipolar disorder, schizophrenia or presence of psychotic symptoms, bulimia nervosa or anorexia nervosa, or current major depressive disorder
* Pregnancy or lactation
* Taking weight loss medications
* Weight change of plus or minus 5% in the last 3 months

Conditions not specifically mentioned above may serve as criteria for exclusion at the discretion of the investigators. Additionally, potential subjects might be excluded if they demonstrate a style of interpersonal relationships that would inhibit successful completion of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2008-09-18 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
The primary goal of the current study is to determine if changes in energy expenditure in response to acute over- and underfeeding are related to variation in changes in weight and body energy stores with longer-term over- and underfeeding. | Ongoing
  Changes in energy expenditure, weight, and body energy stores measured via physical examinations, laboratory studies, questionnaires, body composition assessments, oral glucose tolerance tests, metabolic chamber studies, and free-living energy use studies

SECONDARY OUTCOMES:
Determine if hormones, responses to behavioral testing, adipocyte size, body composition, core temperature, spontaneous activity, and food absorption/excretion are related to changes in EE with over/under-feeding and variation in weight change. | Ongoing
  Changes in hormones, behavior, adipocyte size, body composition, core temperature, spontaneous activity, food absorption/excretion, changes in EE, and weight measured via physical examinations, laboratory studies, questionnaires, body composition assessments, oral glucose tolerance tests, meal tests, activity monitors, metabolic chamber studies, free-living energy use studies, and fat and muscle biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Susanne M Votruba, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Adams M, Montague CT, Prins JB, Holder JC, Smith SA, Sanders L, Digby JE, Sewter CP, Lazar MA, Chatterjee VK, O'Rahilly S. Activators of peroxisome proliferator-activated receptor gamma have depot-specific effects on human preadipocyte differentiation. J Clin Invest. 1997 Dec 15;100(12):3149-53. doi: 10.1172/JCI119870. PMID 9399962
- [Background] Allison DB, Heshka S, Sepulveda D, Heymsfield SB. Counting calories--caveat emptor. JAMA. 1993 Sep 22-29;270(12):1454-6. doi: 10.1001/jama.270.12.1454. PMID 8371446
- [Background] Astrup A, Buemann B, Christensen NJ, Madsen J, Gluud C, Bennett P, Svenstrup B. The contribution of body composition, substrates, and hormones to the variability in energy expenditure and substrate utilization in premenopausal women. J Clin Endocrinol Metab. 1992 Feb;74(2):279-86. doi: 10.1210/jcem.74.2.1530952.
- [Derived] Cabeza de Baca T, Parrington S, Votruba S, Piaggi P, Krakoff J, Chang DC. Adipocyte size, adipose tissue calories, and circulating adipokines, before and after diet-induced weight loss in humans. Endocrine. 2024 May;84(2):490-499. doi: 10.1007/s12020-023-03666-3. Epub 2024 Jan 4. PMID 38172345
- [Derived] Basolo A, Parrington S, Ando T, Hollstein T, Piaggi P, Krakoff J. Procedures for Measuring Excreted and Ingested Calories to Assess Nutrient Absorption Using Bomb Calorimetry. Obesity (Silver Spring). 2020 Dec;28(12):2315-2322. doi: 10.1002/oby.22965. Epub 2020 Oct 7. PMID 33029899
- [Derived] Hollstein T, Basolo A, Ando T, Votruba SB, Walter M, Krakoff J, Piaggi P. Recharacterizing the Metabolic State of Energy Balance in Thrifty and Spendthrift Phenotypes. J Clin Endocrinol Metab. 2020 May 1;105(5):1375-92. doi: 10.1210/clinem/dgaa098. PMID 32118268
- [Derived] Hollstein T, Basolo A, Ando T, Votruba SB, Krakoff J, Piaggi P. Urinary Norepinephrine Is a Metabolic Determinant of 24-Hour Energy Expenditure and Sleeping Metabolic Rate in Adult Humans. J Clin Endocrinol Metab. 2020 Apr 1;105(4):1145-56. doi: 10.1210/clinem/dgaa047. PMID 32002540
- [Derived] Hollstein T, Ando T, Basolo A, Krakoff J, Votruba SB, Piaggi P. Metabolic response to fasting predicts weight gain during low-protein overfeeding in lean men: further evidence for spendthrift and thrifty metabolic phenotypes. Am J Clin Nutr. 2019 Sep 1;110(3):593-604. doi: 10.1093/ajcn/nqz062. PMID 31172178
- [Derived] Piaggi P. Metabolic Determinants of Weight Gain in Humans. Obesity (Silver Spring). 2019 May;27(5):691-699. doi: 10.1002/oby.22456. PMID 31012296
- [Derived] Stinson EJ, Graham AL, Thearle MS, Gluck ME, Krakoff J, Piaggi P. Cognitive dietary restraint, disinhibition, and hunger are associated with 24-h energy expenditure. Int J Obes (Lond). 2019 Jul;43(7):1456-1465. doi: 10.1038/s41366-018-0305-9. Epub 2019 Jan 16. PMID 30651576
- [Derived] Heinitz S, Piaggi P, Yang S, Bonfiglio S, Steel J, Krakoff J, Votruba SB. Response of skeletal muscle UCP2-expression during metabolic adaptation to caloric restriction. Int J Obes (Lond). 2018 Jun;42(5):974-984. doi: 10.1038/s41366-018-0085-2. Epub 2018 May 17. PMID 29777235
- [Derived] Reinhardt M, Thearle MS, Ibrahim M, Hohenadel MG, Bogardus C, Krakoff J, Votruba SB. A Human Thrifty Phenotype Associated With Less Weight Loss During Caloric Restriction. Diabetes. 2015 Aug;64(8):2859-67. doi: 10.2337/db14-1881. Epub 2015 May 11. PMID 25964395